CLINICAL TRIAL: NCT00195533
Title: Monotherapy With Piperacillin-tazobactam Versus Combination Therapy With Piperacillin-tazobactam Plus Glycopeptide as an Initial Empiric Therapy for Fever in Neutropenic Patients. An Observational Prospective Study.
Brief Title: Study Comparing Piperacillin-tazobactam Versus Piperacillin-tazobactam Plus Glycopeptide in Neutropenic Patients
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: PETHEMA (Program for the Study and Treatment of Haematological Malignances) (Unknown)
Other Study IDs: 100943
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Hematological Malignancy; Leukemia; Myelodysplasia; Lymphoma; Myeloma; Stem Cell Transplantation
Keywords: Leukemia; Lymphoma; Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Anemia, Refractory, with Excess of Blasts; Lymphoma; Neoplasms, Plasma Cell | interventions — Piperacillin, Tazobactam Drug Combination; Glycopeptides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood

INTERVENTIONS:
Drug: piperacillin-tazobactam
Drug: glycopeptide

SUMMARY:
The aim of this study is to compare the efficacy and tolerance of piperacillin-tazobactam versus piperacillin-tazobactam plus glycopeptide as initial empiric antibiotic treatment for fever in neutropenic patients. Study of consecutive cohorts(2). First the patients will be included in the monotherapy branch until completing the predicted number of cases. When this happens, the Coordinating Center will communicate it to the participant centers and from then the patients will be included in the combined therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological malignancy or those who had undergone stem cell transplantation for neoplastic disease.
* Fever (>38ºC)
* Neutropenia (absolute neutrophil count < 500 or < 1000 anticipated to fall below 500 cells within 24-48 hours).

Exclusion Criteria:

* Known allergy to any of the antibiotics used in this trial
* A high probability of death within 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematology units
Sampling Method: Non-Probability Sample
Enrollment: 801 (Actual)
Dates: Start 2001-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
- Clinical efficacy evaluation:72 and 96 hours after the initiation of empirical therapy (early evaluation) and at the completion of the therapeutic trial (overall valuation) | 3 months
- Safety evaluation:during the empirical therapy

SECONDARY OUTCOMES:
Microbiological evaluation:at the completion of the therapeutic trial (overall evaluation) | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com
Locations (12):
- Spain (12):
  - A Coruña
  - Alcalá de Henares
  - Alzira
  - Barcelona
  - Castellon
  - Madrid
  - Salamanca
  - Santa Cruz de Tenerife
  - Tarragona
  - Valencia
  - Valladolid
  - Zaragoza